CLINICAL TRIAL: NCT03684343
Title: Comparative Analysis of Filmed Sequences for the Assessment of Discomfort in Atopic Dermatitis of Infants Under 6 Months of Age
Acronym: PRURINEO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulties
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC17.0205 - PRURINEO
Record Dates: First submitted 2018-09-11; First posted 2018-09-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atopic Dermatitis patients (Other): Filmed consultation with a dermatologist. Laterality and tactile sensitivity test.
  Interventions: Other: Filmed consultation with a dermatologist
- Healthy patients (Other): Filmed consultation with a dermatologist. Laterality and tactile sensitivity test.
  Interventions: Other: Filmed consultation with a dermatologist

INTERVENTIONS:
Other: Filmed consultation with a dermatologist — Patient will be seen by a dermatologist for a consultation which will be filmed. During the consult, a laterality test and a tactile sensitivity test will be performed.
  After the consult, videos will be analysed by scientists to identify the frequency of occurrence of each behavior and the percentage of time passed to express each behavior.

SUMMARY:
Atopic dermatitis (AD) is an frequent chronic and itchy inflammatory dermatitis which concern about 20% of pediatric population with a revelation usually toward 3-6 months of live. However, there are very few data about the prevalence of pruritus of young infants and about the discomfort linked with it. While the skin and the nervous system of young infants (Under 6 month) are competent in pruritus experiment, the acquisition of conscious and deliberate motor ability allowing specific scratching of the body parts which are affected is possible only from 6 month. Thus, the diagnosis of AD intensity and the assesment of the potential associated discomfort are hard. At the present time, the diagnosis and the assesment of pruritus of children are based on a hetero-assesment via scales which are not applicable for infants under 6 month. The visual scale "Numeric Rating Scale" validated in adult population seems to be the most specific to assess AD severity. In pediatric population, the use of "Eppendorf Itch Questionnaire" and the american version of "Childhood Atopic Dermatitis Impact Scale" are recommended. Alternatives to clinic and subjective scoring of pruritus severity are described via actigraphy. Thus, a strong statistic correlation have been demonstrated between a nocturne measure of motor activity of wrist, as a reflect of the intensity of pruritus, and infra-red video analysis. But, once again, the technic is not adapted to young infants because of the absence of conscious and oriented motor ability and as a result of less organised sleep/wake cycle.

In order to improve young infants' (Under 6 month) care, the analysis of their behaviours with AD seems to be necessary to better identify a discomfort of these patients.

ELIGIBILITY:
Atopic dermatitis patients :

Inclusion Criteria:

* Young infant Under 6 month
* Patient with AD (SCORAD between 25 and 50 for moderate AD and > 50 for severe AD)
* Informed consent of the patient's parents

Healthy patients :

Inclusion Criteria:

* Young infant under 6 month
* Free of any pathology
* Informed consent of the patient's parents

Exclusion Criteria (for every patients) :

* Acute intercurrent disease
* Severe malformation
* Underage parents or parent unable to give their consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of each behaviors | Day 0
  The frequency of occurrence of each behaviors will be identify.
Percentage of time passed to express each behavior | Day 0
  The percentage of time passed to express each behavior will be noted.

SECONDARY OUTCOMES:
SCORin Atopic Dermatitis | Day 0
  SCORAD is a severity score used for atopic dermatitis. Only patients with AD will performed this test. SCORAD<25 : mild AD; 25<SCORAD<50 : moderate AD and SCORAD >50 : severe AD
Tactile sensitivity test | Day 0
  Von frey filaments will be applied on the patients skin to estimate the reaction threshold to a subtle tactile stimuli.
Laterality test | Day 0
  An object will be presented to the patient and the dermatologist will note the hand used by the patient to take it.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France, France

REFERENCES:
- [Result] Boyard A, Cosnard C, Simon D, Le Pors C, Abasq-Thomas C, Grandgeorge M, Misery L, Henry S, Roue JM. Evidences for gestures associated with pruritus in very young infants: a pilot study. Sci Rep. 2025 Apr 8;15(1):11943. doi: 10.1038/s41598-025-93412-8. PMID 40199912